CLINICAL TRIAL: NCT00745498
Title: Efficacy Study of Pre- and Intra-operative Intravitreal Bevacizumab Injection on Postoperative Vitreous Hemorrhage After Diabetic Vitrectomy
Brief Title: Pre- and Intra-operative Intravitreal Bevacizumab Injection in Diabetic Vitrectomy
Acronym: IBDV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kyu Hyung Park, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-0801-053-004
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Proliferative Diabetic Retinopathy; Vitreous Hemorrhage
Keywords: Proliferative diabetic retinopathy; vitrectomy; bevacizumab; vitreous hemorrhage
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Preop IVB (Experimental): Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) 1 to 14 days before vitrectomy
  Interventions: Drug: Bevacizumab
- Intraop IVB (Experimental): Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) at the end of vitrectomy
  Interventions: Drug: Bevacizumab
- No IVB (No Intervention): Patients will not receive bevacizumab before nor during vitrectomy

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml)
  Other Names: avastin
  Arms: Intraop IVB; Preop IVB

SUMMARY:
The purpose of this study is to determine the effect of pre- and intra-operative bevacizumab injection on postoperative vitreous hemorrhage after diabetic vitrectomy.

DETAILED DESCRIPTION:
Postoperative vitreous hemorrhage(VH) is a common complication after vitrectomy for proliferative diabetic retinopathy. Persistent or recurrent VH can delay visual rehabilitation and give patients much trouble. There have been efforts to lower the incidence of postoperative VH such as using intraoperative gas tamponade and preoperative bevacizumab injection. Bevacizumab(Avastin) is a potent inhibitor of angiogenesis and has been shown to decrease retinal and iris neovascularization in proliferative diabetic retinopathy. Recently there have been reports showing that preoperative intravitreal bevacizumab (IVB) injection could reduce intraoperative bleeding from abnormal vessels and could make surgery easier and more successful.Our hypothesis is that preoperative bevacizumab injection could reduce postoperative VH by way of decreasing the amount of abnormal vessels and intraoperative injection could also reduce postoperative VH by inhibiting the vessel formation after surgery.

To prove our hypothesis, we started the prospective randomized comparative study to determine the effect of pre- and intra-operative IVB injection on postoperative vitreous hemorrhage after diabetic vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first vitrectomy for complications of proliferative diabetic retinopathy such as vitreous hemorrhage, tractional fibrovascular membrane proliferation, tractional or combined retinal detachment)

Exclusion Criteria:

* Follow-up period of less than 6 months
* Intraoperative use of long-acting gas or silicone oil
* Repeat vitrectomy after first vitrectomy for diseases other than vitreous hemorrhage
* Not first vitrectomy
* Uncontrolled hypertension
* Medical history of abnormal blood coagulation
* Time interval between IVB injection and PPV longer than 2 weeks and recent history (within 3 months) of IVB treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Hyung Park, M.D., Principal Investigator — Seoul National Univeristy Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyunggi-do, South Korea

REFERENCES:
- [Background] Chen E, Park CH. Use of intravitreal bevacizumab as a preoperative adjunct for tractional retinal detachment repair in severe proliferative diabetic retinopathy. Retina. 2006 Jul-Aug;26(6):699-700. doi: 10.1097/01.iae.0000225351.87205.69. No abstract available. PMID 16829817

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive diabetic patients requiring pars plana vitrectomy (PPV) for complications of diabetic retinopathy at Seoul National University Bundang Hospital were referred to assess eligibility.
Pre-assignment Details: If indications for PPV included proliferative diabetic retinopathy (PDR) related complications such as nonclearing vitreous hemorrhage (VH), macula-involving or -threatening tractional retinal detachment (TRD) or fibrovascular proliferation with vitreoretinal adhesions, the patient was enrolled in the study.
Groups:
- Preop IVB: Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) 1 to 7 days before vitrectomy
- Introp IVB: Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) at the end of vitrectomy
Period: Overall Study
Arm/Group | Preop IVB | Introp IVB | No IVB
Started | 41 | 43 | 42
Completed | 36 | 37 | 34
Not Completed | 5 | 6 | 8
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Injection of intravitreal silicone oil o | 3 | 4 | 4
Not completed — Non-PDR related VH | 0 | 1 | 1
Not completed — Edophthalmitis after preoperative IVB | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preop IVB | Intraop IVB | No IVB | Total
Number analyzed (Participants) | 41 | 43 | 42 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (9.5) | 55.6 (10.3) | 55.0 (11.4) | 53.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 22 | 57
  Male | 26 | 23 | 20 | 69

OUTCOME MEASURES:

1. Primary Outcome: Recurrent VH Incidence (Early and Late)
Description: Recurrent VH was defined as a new episode of grade 1 or more VH occurring more than 1 week after surgery. "Early recurrent VH" was VH occurring <= 4 weeks and "late recurrent VH" was VH occurring >4 weeks after surgery.
Time Frame: 6 months
Population: With study power of 80%, significance level of 0.05, assumption that IVB injection will decrease postoperative VH incidence from 35% to 10%, a sample size of 40 patients for each group was calculated. The ITT approach was used for analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Preop IVB | Intraop IVB | No IVB
Number analyzed (Participants) | 36 | 37 | 34
Percentage of participants
  Early | 22.2 | 10.8 | 32.4
  Late | 11.1 | 16.2 | 14.7
Statistical Analysis 1: Comparison: Preop IVB vs Intraop IVB vs No IVB; With study power of 80%, a significance level of 0.05, and the assumption that IVB injection will decrease postoperative VH incidence from 35% to 10%, a sample size of 40 patients for each group was calculated; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Secondary Outcome: Initial Time of Vitreous Clearing (ITVC)
Description: The interval in number of days for VH of grade 1 or more observed at postoperative day 1 to clear-up completely. VH of grade 1 was defined as mild vitreous hemorrhage with visible fundus details, but difficult to evaluate the retinal nerve fiber layer or small vessels.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Preop IVB | Intraop IVB | No IVB
Number analyzed (Participants) | 36 | 37 | 34
days | 26.4 (42.5) | 10.3 (8.2) | 25.2 (26.1)

3. Secondary Outcome: Visual Outcome
Description: Best-corrected visual acuity (BCVA) at postoperative 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Preop IVB | Intraop IVB | No IVB
Number analyzed (Participants) | 36 | 37 | 34
logMAR | 0.62 (0.58) | 0.68 (0.47) | 0.51 (0.56)

4. Secondary Outcome: Postoperative Resolution of Neovascularization
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Preop IVB | Intraop IVB | No IVB
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43 | 1/42
Other Adverse Events (participants affected / at risk) | 1/41 | 3/43 | 1/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preop IVB (N=41) | Intraop IVB (N=43) | No IVB (N=42)
Rhegmatogenous retinal detachment immediately following operation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preop IVB (N=41) | Intraop IVB (N=43) | No IVB (N=42)
neovascular glaucoma following surgery (Eye disorders) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No